CLINICAL TRIAL: NCT01465776
Title: A Phase 1b Pilot Study Evaluating Oral Administration of Freeze-Dried Black Raspberries in Pre-Surgical Patients With Oral Squamous Cell Carcinoma
Brief Title: Freeze-Dried Black Raspberries in Treating Patients With Oral Squamous Cell Cancer Undergoing Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amit Agrawal (Other)
Responsible Party: Sponsor-Investigator, Amit Agrawal, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-0497; NCI-2011-02684 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-09-08; First posted 2011-11-07 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Squamous Cell Carcinoma of Mouth
Keywords: SCC of the oral cavity; black raspberries
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemoprevention) (Experimental)
  Interventions: Other: laboratory biomarker analysis; Other: preventative dietary intervention

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies
Other: preventative dietary intervention — lyophilized black raspberries(LBR) administration: 3 LBR troche lozenges (dissolved in mouth), 4 times/day beginning at minimum of 24 hrs following biopsy until night before surgery
  Other Names: dietary; LBR; lyophilized black raspberries

SUMMARY:
This pilot phase I trial studies freeze-dried black raspberries in treating patients with oral squamous cell cancer undergoing surgery. Chemoprevention is the use of certain drugs to keep cancer from forming. Eating freeze-dried black raspberries may help prevent or treat oral cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the relationship between the length of short-term lyophilized black raspberries (LBR) administration to human oral cancer patients and the modulation, in oral cavity tissues, of a subset of specific genes previously identified by us to be "LBR-responsive" and associated with LBR's chemopreventive activity.

SECONDARY OBJECTIVES:

I. To evaluate the effects of LBR administration in humans on cell proliferation, apoptosis, and angiogenesis in oral cavity tissues using various established biomarkers including Ki-67 or proliferating cell nuclear antigen (PCNA), caspase-3, vascular endothelial growth factor (VEGF) or basic fibroblast growth factor (bFGF).

II. To assess the feasibility of administering lyophilized freeze-dried black raspberries in oral troche form to pre-surgical patients diagnosed with squamous cell carcinoma of the oral cavity (compliance, tolerance, adverse events).

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed, biopsy-proven previously untreated squamous cell carcinoma (SCC) of the oral cavity (stages I - IV); suspected cases of SCC will be allowed if biopsy is performed and results of SCC confirmed on subsequent histopathologic analysis (i.e. frozen section) prior to enrollment and initiation of LBR administration
* Patients must already be planned for surgical resection of their tumor (prior to being considered eligible for this study)
* Patients must be able to take nutrition/medications orally
* No prior history of intolerance or allergy to berry or berry-containing products

Exclusion Criteria:

* History of intolerance (including hypersensitivity or allergy) to berry or berry-containing products
* Known history of bleeding disorder or patient on systemic anticoagulation therapy (i.e. coumadin, heparin) for purposes of the study biopsy
* Pregnant women; although there are no known adverse effects of black raspberries upon the fetus, if patients become pregnant during period of LBR administration, then LBR will be discontinued and patient will be removed from the study
* Inability to grant informed consent
* Patients must not be planning to receive chemotherapy or radiation therapy prior to their surgery or this will affect endpoint analysis and these patients will be excluded from the study
* Patients taking cyclooxygenase (COX)-I or COX-2 inhibitors, who cannot be taken off the medication due to their clinical condition will be excluded given that these agents may interfere with biomarkers studied
* Vegetarians will be excluded from the study since we anticipate that this patient population will have difficulty adhering to a low-phenolic diet (restricts basically all plant-based foods)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-01-10 (Actual); Primary Completion 2010-02-16 (Actual); Study Completion 2010-02-16 (Actual)

PRIMARY OUTCOMES:
Relationship between the length of short-term LBR administration to human oral cancer patients and the modulation, in oral cavity tissues, of LBR-responsive genes | up to 60 months
  Statistical summaries of biopsy to surgery changes in quantitative real-time RT-PCR data made on the log scale (geometric mean of percent changes +/- s.e. expressed as a percentage).Confidence intervals produced and significance of the correlation between real-time RT-PCR values and period of treatment (i.e. time from biopsy to surgery) using Fisher's transformation of Spearman's rank correlation tested. Semi-quantitative IHC analyzed using an ordinal logistic model to determine significance of associations between period of treatment and change in staining from biopsy to surgery.

SECONDARY OUTCOMES:
Evaluate effects of lyophilized freeze-dried black raspberries (LBR) administration in humans on cell proliferation, apoptosis, and angiogenesis in oral cavity tissues using various established biomarkers. | up to 60 months
  Biomarkers include Ki-67, PCNA, caspase-3, VEGF, or bFGF
Assess feasibility of administering lyophilized freeze-dried black raspberries in oral troche form to pre-surgical patients diagnosed with squamous cell carcinoma of the oral cavity. | from 7-28 days

CONTACTS AND LOCATIONS:
Overall Officials: Amit Agrawal, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Background] Knobloch TJ, Uhrig LK, Pearl DK, Casto BC, Warner BM, Clinton SK, Sardo-Molmenti CL, Ferguson JM, Daly BT, Riedl K, Schwartz SJ, Vodovotz Y, Buchta AJ Sr, Schuller DE, Ozer E, Agrawal A, Weghorst CM. Suppression of Proinflammatory and Prosurvival Biomarkers in Oral Cancer Patients Consuming a Black Raspberry Phytochemical-Rich Troche. Cancer Prev Res (Phila). 2016 Feb;9(2):159-71. doi: 10.1158/1940-6207.CAPR-15-0187. Epub 2015 Dec 23. PMID 26701664
- See also: Jamesline — http://cancer.osu.edu